CLINICAL TRIAL: NCT03120065
Title: Virologic Treatment Failure and Drug Resistance in HIV-infected Kenyan Children
Brief Title: Virologic Treatment Failure and Drug Resistance in HIV-infected Kenyan Children (RESPECT)
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Vreeman, MD, MS (Other)
Collaborators: Moi University (Other); Brown University (Other)
Responsible Party: Sponsor-Investigator, Rachel Vreeman, MD, MS, Associate Professor, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1601396087
Record Dates: First submitted 2017-03-06; First posted 2017-04-19 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Viral Resistance; Treatment Failure
Keywords: adherence
MeSH Terms: interventions — Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEMS follow up (Other): Approximately 25% of the enrolled study population will have their adherence to medicines monitored by research personnel through the use of electronic dose monitoring caps (MEMS) for a period of 3 months. The participant's ART medication regimen will be dispensed in a bottle with a cap that monitors the time and date in which the cap is opened. Each month, the participant will bring the bottle with them on their clinic day for three months and the research personnel will extract the timing information from the cap.
  Interventions: Other: Electronic Dose Monitoring (MEMS)

INTERVENTIONS:
Other: Electronic Dose Monitoring (MEMS) — The MEMS cap is an electronic bottle cap that records the time and date of a bottle being opened. The research personnel will extract the timing of the MEMS bottle opening events for adherence analysis.

SUMMARY:
The primary objective of this study is to use a well-characterized pediatric AMPATH cohort, with detailed medication-taking, drug level, and clinical data, to longitudinally evaluate treatment failure and drug resistance to improve long-term care for HIV-infected children in Kenya and other RLS. Examining treatment failure and drug resistance emergence in children on ART and what factors impact these negative outcomes, will provide needed data to critically evaluate the efficacy of current ART, weight-based pediatric drug dosing guidelines, and recommendations for subsequent therapies. The objective is to specifically characterize how non-adherence leads to a lack of viral suppression and to drug resistance evolution, and how this characterization can inform interventions to improve adherence and increase treatment success.

DETAILED DESCRIPTION:
Resistance to antiretroviral therapy (ART) hampers effective treatment of pediatric HIV infection and can undermine long-term clinical care outcomes. In resource-limited settings (RLS), where 90% of the world's HIV-infected children live, the risk and impact of ART failure and resistance development are particularly significant due to limited treatment monitoring, restricted medication options and lifelong ART needs, from birth through adolescence and into adulthood. Children in RLS therefore face serious clinical consequences when their virus is not suppressed, but few longitudinal data are available to inform pediatric clinical guidelines or direct interventions to minimize those risks. How specific patterns of medication non-adherence or challenges with appropriate ART dosing might impact ART failure and the development of drug resistance are poorly understood for children in RLS. The primary objective of this study is to use a well-characterized pediatric AMPATH cohort, with detailed medication-taking, drug level, and clinical data, to longitudinally evaluate treatment failure and drug resistance to improve long-term care for HIV-infected children in Kenya and other RLS. Examining treatment failure and drug resistance emergence in children on ART and what factors impact these negative outcomes, will provide needed data to critically evaluate the efficacy of current ART, weight-based pediatric drug dosing guidelines, and recommendations for subsequent therapies. The objective is to specifically characterize how non-adherence leads to a lack of viral suppression and to drug resistance evolution, and how this characterization can inform interventions to improve adherence and increase treatment success. AMPATH cares for over 80,000 adult and pediatric HIV-infected patients in western Kenya, including over 2,800 children on ART.

The research objective of this application will be accomplished by pursuing the following five specific aims: Aim 1: Determine prevalence of viral failure and examine resistance mutations among a retrospective study cohort of 685 perinatally HIV-infected Kenyan children on 1st-line ART; Aim 2: Investigate associations between specific adherence patterns, ART drug levels and other demographic and clinical factors, with viral failure and drug resistance; Aim 3: Study long-term immunologic, virologic and drug resistance outcomes and their associations in prospectively re-enrolled study participants; Aim 4: Enhance analyses of viral failure, drug resistance accumulation and associated demographic and clinical factors by examining the longitudinal banked samples available for a subset of the study cohort (n=327); Aim 5: Develop a data-driven intervention algorithm to identify children at risk for viral failure and resistance.

The hypothesis of this study proposes that there will be high levels of treatment failure and drug resistance associated with patterns of non-adherence and inadequate drug levels.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in CAMP study
* Viable banked blood sample; HIV-infected documented by DNA-PCR (Amplicor, Roche, Basel, Switzerland) for children less than 18 months of age and by 2 parallel HIV rapid ELISA tests using Determine and Bioline for children older than 18 months of age.
* < 19 years of age

Exclusion Criteria:

Mental or physical incapacity of legal caregiver leading to inability to provide informed consent

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 499 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Viral Resistance | 18 months
  Blood samples will be analyzed for viral resistance testing, both for retrospective and prospective samples samples (TP1)

SECONDARY OUTCOMES:
Adherence MEMS | 3 months
  Adherence will be monitored via MEMS bottle caps
Adherence CAMP | 3 months
  Adherence will be assessed via CAMP questionnaire
Clinical Data: WHO stage | 6 years
  WHO stage will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Viral Load | 6 years
  Longitudinal viral loads will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Weight | 6 years
  Longitudinal weight will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Height | 6 years
  Longitudinal height will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Regimen | 6 years
  Longitudinal regimen will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Opportunistic Infections | 6 years
  Longitudinal opportunistic infections will be analyzed for associations with viral resistance and treatment failure in this cohort.
Clinical Data: Disclosure Status | 6 years
  Longitudinal disclosure status will be analyzed for associations with viral resistance and treatment failure in this cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C Vreeman, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Moi Teaching and Referral Hospital - AMPATH Center, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No